CLINICAL TRIAL: NCT05071495
Title: TeleDiet Study: A Randomized Controlled Study Investigating the Impact of Dietary Education and Counseling With a Smartphone Application on Secondary Prevention of Coronary Artery Disease
Brief Title: TeleDiet Study: The Impact of Dietary Education and Counseling With a Smartphone Application on Secondary Prevention of Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/171
Record Dates: First submitted 2021-09-13; First posted 2021-10-08 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Secondary Prevention; Diet Therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: Smartphone application
- Control group (No Intervention)

INTERVENTIONS:
Device: Smartphone application — Smartphone application named "Signal", which connects patients and health providers
  Arms: Intervention group

SUMMARY:
Digital cardiology is gaining power in the field of preventive cardiology recently, and several trials have already shown good results of dietary therapy with digital cardiology. However, there has been no reports that showed effect of dietary counseling through digital cardiology for secondary prevention of coronary artery disease.

TeleDiet study investigates the impact of dietary therapy with a smartphone application on the content of meals and metabolic parameters for patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Owning a smartphone and able to use it
2. Written informed consent obtained
3. Starting cardiac rehabilitation
4. Coronary artery disease

Exclusion Criteria:

1. Special diet due to other reasons (eg. renal diet, pancreatic insufficiency diet)
2. Age <18 years old
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
MedDiet score (the Mediterranean diet score) | Up to 3 months
  This score has the extreme values of 0 (minimum) and 55 (maximum). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Blood lipid tests (LDL-cholesterol [LDL-C], HDL-cholesterol [HDL-C], and triglyceride [TG]) | Up to 3 months
Blood glycated hemoglobin (HbA1c) test | Up to 3 months
Blood creatinine (Cr) test | Up to 3 months
Parameters in the ergospirometer test (maximal oxygen consumption [VO2 max]) | Up to 3 months
Parameters in the ergospirometer test (anaerobic threshold [AT]) | Up to 3 months
Values of self-efficacy (questionnaire of General Self-Efficacy Scale [GSE]) | Up to 3 months
  This scale has the extreme values of 10 (minimum) and 40 (maximum). Higher scores mean a better outcome.
Values of medication adherence (questionnaire of Identification of Medication Adherence Barriers [IMAB]) | Up to 3 months
  This scale has the extreme values of 30 (minimum) and 150 (maximum). Higher scores mean a worse outcome.
Values of quality of life (Health-related Quality of Life questionnaire [HeartQoL]) | Up to 3 months
  This scale has the extreme values of 0 (minimum) and 42 (maximum). Higher scores mean a better outcome.
Body weight (BW) | Up to 3 months
Body mass index (BMI) | Up to 3 months
  Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, Principal Investigator — Jessa Ziekenhuis vzw
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium